CLINICAL TRIAL: NCT05475743
Title: Early Effects of a Pain Informed Movement Program in Patients With Post COVID-19 Condition Experiencing Persistent Pain: a Randomized Control Trial
Brief Title: Pain Informed Movement Program in Patients With Post COVID-19 Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0097UG
Record Dates: First submitted 2022-07-26; First posted 2022-07-27 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Informed Movement program (Experimental)
  Interventions: Other: Pain Informed Movement program
- Standard medical care and leaflet education (Active Comparator)
  Interventions: Other: Standard medical care and leaflet education

INTERVENTIONS:
Other: Pain Informed Movement program — The patients included in the experimental group attended an 8-week Pain Informed Movement program in addition to standard medical care. The program was led by a physical therapist with experience in treating patients with chronic pain. This program consisted of 2 face-to-face sessions per week, and they were asked to complete two sessions at home weekly. The first face-to-face session was a group session with 3-6 participants, and the second face-to-face session was individual. Both sessions lasted approximately 1 h. In the group sessions, pain neuroscience education was conducted. In the individual sessions, an individualized functional exercise program was performed by each patient, as well as relaxation techniques. Patients were asked to perform the functional exercises and relaxation techniques at home. Participants were asked to record their compliance with the program and their progress.
  Arms: Pain Informed Movement program
Other: Standard medical care and leaflet education — In addition to standard medical care, patients assigned to this group received a leaflet with information about the main post COVID-19 condition symptoms. This is a control group that was not controlled or monitored by a therapist.
  Arms: Standard medical care and leaflet education

SUMMARY:
Patients who have undergone COVID-19 infection often have long-term sequelae. One of the most prevalent sequelae is pain. The main objective of this research is to investigate the efficacy of Pain Informed Movement program in patients with post COVID-19 condition experiencing persistent pain. Through the implementation of this program, the investigators seek to determine whether such intervention can offer significant improvements in reducing pain intensity and interference, catastrophizing, kinesiophobia, and functionality of affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Agreed to participate.
* Post COVID-19 condition patients meeting the WHO definition for this disease.
* Patients with moderate or severe pain were included, the cut-off point on the Visual Analogical Scale (VAS) being pain greater than or equal to 3.5 cm.

Exclusion Criteria:

* Pulmonary, cardiac, neurological, vascular, or orthopaedic pathologies that could limit the execution of the evaluation and intervention.
* Cognitive impairment that prevented them from understanding and answering the questionnaires.
* Patients suffering from a reinfection with SARS-CoV-2.
* Patients with a history of severe or critical COVID-19 disease severity.
* Patients who had pre-existing chronic pain according to the current IASP definition.
* Patients participating in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity and pain interference | Baseline and at 8 weeks at the end of the intervention
  Pain intensity and interference were quantified using the Brief Pain Inventory (BPI). The section intended to measure pain intensity on the BPI comprises four items, while the section related to pain interference includes seven items. In the intensity section, responses range on a scale from 0 (no pain) to 10 (maximum pain), while in the interference section, responses range from 0 (no interference) to 10 (total interference). To calculate the severity and interference index, the values of the corresponding items are averaged, obtaining values ranging from 0 to 10, with a higher score indicating greater pain intensity and interference. The BPI has been validated as a reliable and valid tool to evaluate these aspects of pain.
Changes in catastrophization | Baseline and at 8 weeks at the end of the intervention
  To evaluate the phenomenon of catastrophizing, the Pain Catastrophizing Scale (PCS) was applied. This instrument consists of 13 statements structured on a 5-point Likert scale ranging from 0 (at no time) to 4 (at all times). The PCS breaks down catastrophizing into three components: feelings of helplessness, magnification of difficulties, and rumination about pain. Each of the items describes different thoughts and emotions that people may experience when in pain. The final score is obtained by summing the scores of all the items, resulting in a score ranging from 0 to 52, with higher scores indicating a higher level of catastrophizing.
Changes in kinesiophobia | Baseline and at 8 weeks at the end of the intervention
  The Tampa Kinesiophobia Scale (TSK) was used to quantify apprehension related to physical activity and the fear of injury (or re-injury). This scale is composed of 11 statements, which are assigned a score on a 4-point scale (1-4). Total scores vary between 11 and 44 points, with higher values being indicative of greater fear of movement and the possibility of (re)injury.
Changes in functionality | Baseline and at 8 weeks at the end of the intervention
  Functionality was assessed using the WHODAS 2.0 tool (World Health Organization Disability Assessment Schedule). It consists in 36 items assessing six main areas of functional ability. This questionnaire uses a 5-point Likert scale for respondents to rate their level of difficulty in six main subscales: Cognition, Mobility, Self-Care, Interpersonal Relationships, Home Life and Community Involvement. Response options go from 1 (no difficulty) to 5 (extreme difficulty or can not do). The scores obtained in each area are added to obtain a total score that shows the degree of functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain